CLINICAL TRIAL: NCT03688243
Title: Non Exudative Age-Related Macular Degeneration Imaged With Swept Source Optical Coherence Tomography
Brief Title: Non Exudative AMD Imaged With SS-OCT
Acronym: BIRC-01
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston Image Reading Center (Industry)
Responsible Party: Sponsor
Other Study IDs: BIRC-01 IMPACT; NCT03972800 (obsolete NCT alias)
Record Dates: First submitted 2018-09-25; First posted 2018-09-28 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Dry Macular Degeneration
Keywords: AMD; early AMD; intermediate AMD; Geographic Atrophy; nascent GA
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At baseline or follow up, an optional blood sample for future exploratory genetics analysis will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Cohort 1 'IMPACT Cohort': Subjects with intermediate AMD in both eyes, and at least one eye with a drusen volume in the central 3 mm circle centered on the fovea of at least 0.02mm3 in the absence of GA or nGA as diagnosed with OCT en face imaging OR subjects with AMD (early or intermediate) diagnosed in one eye and exudative AMD diagnosed in the fellow eye will undergo SS-OCT imaging every 3 months for 2 years
  Interventions: Device: SS-OCT imaging
- Cohort 2 'SWAGGER Cohort': Subjects with GA or nGA secondary to AMD that is at least the size of a large druse (125 microns in diameter; 0.05 mm2) and no greater than 7 disc areas (17 mm2) in at least one eye will undergo SS-OCT imaging every 3 months for 2 years
  Interventions: Device: SS-OCT imaging
- Cohort 3: Subjects with GA enrolled in another trial
  Interventions: Device: SS-OCT imaging

INTERVENTIONS:
Device: SS-OCT imaging — All subjects will undergo retinal imaging using the Zeiss PlexElite SS-OCT, a non-contact, non-invasive ocular imaging instrument
  Other Names: Zeiss PlexElite; PlexElite 9000; Swept Source OCT; Optical Coherence Tomography Angiography

SUMMARY:
The investigators wish to better understand the role of the choriocapillaris (CC) in the formation and progression of non-exudative in age related macular degeneration (armd) by imaging the retinal pigment epithelium (rpe) and the choroidal microvasculature and by studying their inter-dependence to determine if the loss of the CC could prove useful as an anatomic clinical trial endpoint in future drug trials.

DETAILED DESCRIPTION:
This is a longitudinal observational study where the investigators will look at 450 subjects, 200 with intermediate AMD in at least one eye, or with AMD in one eye, either early or intermediate, and with late AMD (exudative) in the other eye, and 250 subjects with nGA or GA in at least one eye.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 and over
2. Clinic diagnosis of non-exudative iAMD in at least one eye with a drusen volume in the central 3 mm circle centered on the fovea of at least 0.02 mm3 in the absence of GA or nGA as diagnosed with OCT en face imaging OR Clinical diagnosis of early or early/intermediate stage AMD in one eye in the absence of nGA or GA and exudative AMD in the other eye OR clinical diagnosis of GA or nGA secondary to AMD that is at least the size of a large druse (125 microns in diameter; 0.05 mm2) and no greater than 7 disc areas (17 mm2) in at least one eye which has never been treated with anti-VEGF agents
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from the study:

1. Below the age of 50
2. Subjects with exudative AMD in both eyes
3. Eyes with evidence of non-proliferative and proliferative diabetic retinopathy.
4. Presence of confounding ocular diagnosis such as myopia >6D, or other ocular conditions that may cause retinal pigment epithelium atrophy or exudative MNV
5. Subjects unable to give informed consent.
6. Subjects who are unable to comply with imaging guidelines

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with intermediate AMD, Geographic Atrophy and nascent Geographic Atrophy.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in Choroidal Perfusion Deficits at 1 year compared to Baseline | 1 year time point
  Assessment of Choriocapillaris perfusion

SECONDARY OUTCOMES:
Pre-existing sub-clinical Macular Neovascularization (MNV) | 1 year and 2-year time points
  Presence of abnormal new vessels arising from the Choroid
Automated Drusen Volume measurements | 1 year and 2-year time points
  Compare the automated measurements of drusen volume using the Zeiss algorithm with manual measurements by trained readers
Automated GA measurements | 1 year and 2-year time points
  Compare the automated measurements of GA area using the Zeiss algorithm with manual measurements by trained readers
Structural OCT markers and Genetic Markers | 1 year and 2-year time points
  Correlate structural markers on SS-OCT/OCTA with genetic markers of disease

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Waheed, MD, Principal Investigator — Boston Image Reading Center/Tufts Medical Center; Philip Rosenfield, MD, PhD, Principal Investigator — Bascom Palmer Eye Institute
Locations (5):
- United States (4):
  - University of California Los Angeles Doheny Eye Institute, Los Angeles, California
  - Bascom Palmer Eye Institue, Miami, Florida
  - New England Eye Center/Tufts Medical Center, Boston, Massachusetts
  - Vitreous Retina Macular Consultants of NY, New York, New York
- Melbourne University CERA, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided